CLINICAL TRIAL: NCT06175260
Title: Investigation on the Efficacy of Oral Carnitine Challenge Test Based on a Gut Microbiota Functional Test
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201906010RINC
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2019-06

CONDITIONS: Dysbiosis; Healthy
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from fecal samples were extracted and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: oral carnitine challenge test — Urine samples will be collected to quantify trimethylamine N-oxide (TMAO) levels at four time points: before, and 24, 48, and 72 hours after the oral administration of 1500 mg of L-carnitine.

SUMMARY:
This study seeks to enlist healthy volunteers to form a validation cohort. The purpose is to confirm the observed correlations between the gut microbiome and the capacity to produce trimethylamine N-oxide (TMAO), which will be assessed using the oral carnitine challenge test (OCCT).

DETAILED DESCRIPTION:
Carnitine, a nutrient widely found in meat, can promote the use of fatty acids by mitochondria to produce energy in the human body. It was previously thought to be beneficial in helping the body consume fat for energy and might be helpful for muscle training or weight loss. However, some human populations have harmful bacteria in their intestines that compete with the body for the use of carnitine. These bacteria metabolize carnitine to produce potentially harmful Trimethylamine N-oxide (TMAO). This might be one of the reasons why long-term consumption of red meat, which is rich in carnitine, is associated with a higher risk of cardiovascular disease. Therefore, understanding the functional state of one's gut microbiota and whether it is suitable to consume foods rich in carnitine can greatly aid in long-term dietary and health planning. In recent years, we have established an oral carnitine challenge test that (OCCT) can distinguish whether the intestinal bacteria in a subject produce a large amount of TMAO in the body. This was published in the Gut journal in 2019 and is expected to provide dietary or nutritional supplement recommendations for personalized nutrition for the test subjects. However, the value of the carnitine challenge test in distinguishing between high TMAO producers and low TMAO producers, and whether it can serve as an effective reference for whether a subject is suitable to consume large amounts of meat or take carnitine supplements, still needs further experimental verification. This study seeks to enlist healthy volunteers to form a validation cohort. The purpose is to confirm the observed correlations between the gut microbiome and the capacity to produce TMAO, which will be assessed using the OCCT.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 20 and above who are willing to participate in the trial.

Exclusion Criteria:

1. Under the age of 20
2. History of gastrointestinal surgery
3. History of malignant tumors
4. Those who have used antibiotics, probiotics, or carnitine supplements within the past month will be excluded
5. Liver cirrhosis
6. End-stage kidney disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals undergoing health examinations at the Health Management Center of National Taiwan University Hospital.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Trimethylamine N-oxide (TMAO) production capacity measured by oral carnitine challenge test (OCCT) | at enrollment
  The area under the curve of TMAO levels under OCCT

SECONDARY OUTCOMES:
Correlations between the gut microbiome and the capacity to produce TMAO | at enrollment
  The gut microbiome indicated microbial genes and taxonomies measured by shotgun metagenome sequencing whereas TMAO producing capacity was measured by OCCT.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided